CLINICAL TRIAL: NCT04410042
Title: Tranexamic Acid (TXA) to Reduce Volume Of Blood Transfused In Pediatric And Young Adult Cancer Patients Undergoing Limb Salvage Procedure Of A Lower Extremity
Brief Title: Tranexamic Acid Use to Reduce Blood Transfusion in Pediatric Cancer Patients Undergoing Limb Salvage Procedure
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Per sponsor
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: TXAKIDS; NCI-2020-02984 (Registry Identifier: NCI Clinical Trial Registration Program)
Record Dates: First submitted 2020-05-08; First posted 2020-06-01 (Actual); Results first posted 2024-12-05 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Cancer of the Bone; Limb Salvage
Keywords: Blood Transfusion; Cancer of the bone; Distal femur; Limb Salvage; Malignant Bone Tumor; Placebo; Proximal tibia; Randomized; Tranexamic acid; TXA
MeSH Terms: conditions — Bone Neoplasms | interventions — Tranexamic Acid; Sodium Chloride; Fluoridation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: To allow for the study team and participants to remain blinded to the treatment assignment, the study drug will be labeled as Tranexamic Acid/Placebo (TXAKIDS) followed by applicable dose and administration instructions.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Tranexamic Acid (Experimental): At initiation of surgical preparation, participants randomized to the active treatment arm will receive tranexamic acid 10 mg/kg (max 1 g), given via syringe pump programmed to infuse over 15 minutes. If no unacceptable toxicities occur, a second dose of tranexamic acid IV push over 5 to 15 minutes will be given 6 hours (with a window of +/- 30 minutes) after the first dose (either intra- or post-operatively).
  Interventions: Drug: Tranexamic Acid
- Placebo (Placebo Comparator): At initiation of surgical preparation, participants randomized to the placebo treatment arm will receive 0.9% sodium chloride (salt water). It will be matched in appearance, volume, and administration to the active treatment arm with tranexamic acid. If no unacceptable toxicities occur, a second dose of placebo IV push over 5 to 15 minutes will be given 6 hours (with a window of +/- 30 minutes) after the first dose (either intra- or post-operatively).
  Interventions: Other: 0.9% sodium chloride

INTERVENTIONS:
Drug: Tranexamic Acid — Given IV
  Other Names: Cyklokapron®
  Arms: Tranexamic Acid
Other: 0.9% sodium chloride — Given IV
  Other Names: Salt water
  Arms: Placebo

SUMMARY:
This is a randomized double-blind control trial evaluating the use Tranexamic acid (TXA) to decrease blood loss and transfusion requirements in pediatric and young adult cancer patients undergoing a limb salvage procedure that frequently requires perioperative or post-operative transfusions of blood products.

Primary Objective

* To evaluate the difference in intra-or post-operatively transfused blood volume (mL/kg) for patients undergoing limb salvage procedures of the distal femur or proximal tibia who are randomized to receive perioperative tranexamic acid (TXA) versus placebo.

Secondary Objectives

* To evaluate changes in platelets and in hemoglobin from pre-op to post-op level for patients randomized to receive perioperative TXA versus placebo.
* To evaluate differences in post-operative daily surgical drain output for patients randomized to receive perioperative TXA versus placebo.
* To evaluate changes in estimated blood loss (EBL) for patients randomized to receive perioperative TXA versus placebo.
* To evaluate the association between the intra-or post-operatively transfused blood volume and estimated blood loss (EBL) for patients randomized to receive perioperative TXA and placebo, respectively.

Exploratory Objectives

* To evaluate differences in functional outcomes post-operatively for patients randomized to receive perioperative TXA versus placebo.
* To explore if significant correlations are observed between parameters reported with rotational thromboelastometry (ROTEM®) and EBL and transfusion requirements in pediatric and young adult patients undergoing limb salvage procedure who are randomized to perioperative TXA versus placebo.
* To evaluate differences in the prevalence and management of wound complications such as superficial or periprosthetic infections, wound dehiscence, contact dermatitis, post- operative hematomas, or any other clinically significant wound complication between patients randomized to receive perioperative TXA versus placebo.

DETAILED DESCRIPTION:
Eligible participants undergoing limb salvage procedures will be randomized to receive either tranexamic acid (TXA) or placebo peri-operatively.

The initial dose of tranexamic acid/placebo will be given at the initiation of surgical preparation. The second dose will be given 6 hours after the first dose (either intraoperatively or post-operatively). All doses will be given intravenously. Doses will be double blinded and randomized for each surgical procedure.

ELIGIBILITY:
Inclusion Criteria:

* Participant undergoing limb salvage procedure of malignant bone tumor of the distal femur or proximal tibia, which typically requires blood transfusions.
* Patient under the age of 25
* Adequate bone marrow function defined as:

  * Upward trending peripheral absolute neutrophil count (ANC)
  * Platelet count ≥ 100,000/mm^3 (transfusion independent defined as no platelets required for 4 days)
  * Hemoglobin ≥ 8.0 g/dL
  * No RBC transfusion within 24 hours
* Adequate renal function defined as:

  * Creatinine clearance or radioisotope GFR ≥ 70 mL/min/1.73m^2 OR
  * Maximum serum creatinine based on age/gender as follows: Age 1 day to < 1 years: maximum serum creatinine (mg/dL) 0.6 for males and 0.5 for females; Age 1 to < 2 years: maximum serum creatinine (mg/dL) 0.6 for males and 0.6 for females; Age 2 to < 6 years: maximum serum creatinine (mg/dL) 0.8 for males and 0.8 for females; Age 6 to < 10 years: maximum serum creatinine (mg/dL) 1.0 for males and 1.0 for females; Age 10 to < 13 years: maximum serum creatinine (mg/dL) 1.2 for males and 1.2 for females; Age 13 to < 16 years: maximum serum creatinine (mg/dL) 1.5 for males and 1.4 for females; Age ≥ 16 years: maximum serum creatinine (mg/dL) 1.7 for males and 1.4 for females
* Adequate liver function defined as:

  * Total bilirubin ≤ 1.5x the institutional upper limit of normal (IULN) for age
  * ALT (SGPT) and AST (SGOT) ≤ 2.5x IULN for age (or <5x IULN for patients with documented disease involving the liver or 10x IULN for patients receiving HDMTX)
  * Serum albumin > 2 g/dL
* Adequate coagulation function as defined by International Normalized Ratio (INR) ≤ 1.5
* Female participants of child-bearing potential (>10 years old) must have a negative serum or urine pregnancy test within 72 hours of sedation

Exclusion Criteria:

* Participants whose limb salvage procedure may require significant manipulation of major blood vessels.
* Participants with known bone marrow deficiency resulting in red blood cell deficiency (e.g. Diamond-Blackfan anemia)
* Participants receiving erythropoietin-stimulating agents (e.g. epoetin alfa)
* Participants with active hemorrhagic cystitis (e.g. alkylator-induced) with gross hematuria or >50 RBCs per high powered field on urinalysis
* Participants actively receiving all-trans retinoic acid (ATRA) or isotretinoin (Accutane)
* Participants with known allergies to antifibrinolytics
* Participants with known hypercoagulopathies
* Personal history of a thrombosis or active thrombus
* Participants currently on anticoagulation medications (e.g. warfarin, enoxaparin)
* Participants with a history of seizures. Patients with a history of febrile seizure are eligible.
* Persisting toxicity related to other systemic therapies (e.g. chemotherapy) which constitutes an unacceptable safety risk based on the judgment of the PI and/or the primary treating physician.
* Female participants who are currently pregnant or actively breastfeeding.
* Female participants who are currently receiving estrogen-based contraception therapy.
* Inability or unwillingness of research participant or legal guardian/representative to give written informed consent.
* Participants enrolled in another clinical trial utilizing an IND/IDE experimental therapy.
* Participants with a history of CNS disease.
* Participants with known bleeding disorder.
* Participants with known platelet dysfunction.

Max Age: 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Actual)
Dates: Start 2021-01-29 (Actual); Primary Completion 2024-01-16 (Actual); Study Completion 2024-01-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael D. Neel, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant de-identified datasets containing the variables analyzed in the published article will be made available (related to the study primary or secondary objectives contained in the publication). Supporting documents such as the protocol, statistical analyses plan, and informed consent are available through the CTG website for the specific study. Data used to generate the published article will be made available at the time of article publication. Investigators who seek access to individual level de-identified data will contact the computing team in the Department of Biostatistics (ClinTrialDataRequest@stjude.org) who will respond to the data request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be made available at the time of article publication.
Access Criteria: Data will be provided to researchers following a formal request with the following information: full name of requestor, affiliation, data set requested, and timing of when data is needed. As an informational point, the lead statistician and study principal investigator will be informed that primary results datasets have been requested.

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: ClinicalTrials Open at St. Jude — http://www.stjude.org/protocols

RESULTS

PARTICIPANT FLOW:
Recruitment Details: As of the data freeze date (12/14/2023), 15 patients are enrolled and 13 of them are eligible. The ineligible reason for one patient is ANC did not meet eligible levels prior to surgery. The second ineligible patient was found to be on oral estrogen contraception after receiving study drug and undergoing surgery. One patient was consented, then consent was withdrawn prior to any study procedures. This patient was not randomized.
Groups:
- Arm A-Tranexamic Acid: At initiation of surgical preparation, participants randomized to the active treatment arm will receive tranexamic acid 10 mg/kg (max 1 g), given via syringe pump programmed to infuse over 15 minutes. If no unacceptable toxicities occur, a second dose of tranexamic acid IV push over 5 to 15 minutes will be given 6 hours (with a window of +/- 30 minutes) after the first dose (either intra- or post-operatively).
  Tranexamic Acid: Given IV
- Arm B-Placebo: At initiation of surgical preparation, participants randomized to the placebo treatment arm will receive 0.9% sodium chloride (salt water). It will be matched in appearance, volume, and administration to the active treatment arm with tranexamic acid. If no unacceptable toxicities occur, a second dose of placebo IV push over 5 to 15 minutes will be given 6 hours (with a window of +/- 30 minutes) after the first dose (either intra- or post-operatively).
  0.9% sodium chloride: Given IV
Period: Overall Study
Arm/Group | Arm A-Tranexamic Acid | Arm B-Placebo
Started | 7 | 7
Completed | 6 | 6
Not Completed | 1 | 1
Not completed — Not Eligible | 1 | 1

BASELINE CHARACTERISTICS:
Population: Eligible participants undergoing limb salvage procedures will be randomized to receive either TXA or placebo peri-operatively - one dose at initiation of surgical preparation and a second dose 6 hours after the first.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A-Tranexamic Acid | Arm B-Placebo | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 16.40 (2.47) | 13.77 (3.25) | 15.08 (3.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 5
  Male | 4 | 3 | 7
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 5 | 5 | 10
  Asian | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: To Evaluate the Difference in intra-or Post-operatively Transfused Blood Volume (mL/kg) for Patients Undergoing Limb Salvage Procedures of the Distal Femur or Proximal Tibia Who Are Randomized to Receive Perioperative Tranexamic Acid (TXA) Versus Placebo.
Description: The intra-or post-operative volumes of transfused blood for both the TXA treated group and placebo group will be estimated with a two-sided 95% confidence interval. The blood volumes transfused per kilogram of body weight of the two groups (TXA vs. Placebo) will be evaluated using a two-sided student's t-test after log(1+x) transformation.
Time Frame: intra- or post-operatively transfused blood volume (mL/kg), 6 months
Measure: Mean (Standard Deviation); unit: mL/kg
Groups:
- TXAKIDS: Eligible participants undergoing limb salvage procedures will be randomized to receive either TXA or placebo peri-operatively - one dose at initiation of surgical preparation and a second dose 6 hours after the first.
Arm/Group | Arm A-Tranexamic Acid | Arm B-Placebo | TXAKIDS
Number analyzed (Participants) | 6 | 6 | 12
mL/kg
  Transfused blood volume, intra-operative (intra-op) | 5.04 (2.34) | 5.15 (2.85) | 5.12 (2.51)
  Transfused blood volume, post-operative (post-op) | 5.74 (1.79) | 5.64 (2.06) | 5.71 (1.85)
Statistical Analysis 1: Comparison: Arm A-Tranexamic Acid vs Arm B-Placebo; Test type: Equivalence — Two-sided test at 0.05 level; p = 0.4000, Wilcoxon rank sum test

2. Secondary Outcome: To Evaluate Changes in Platelets From Pre-op to Post-op Level for Patients Randomized to Receive Perioperative TXA Versus Placebo.
Description: Summary statistics will be provided for the changes in platelet level for both the TXA and placebo group. Two sample t-test or Wilcoxon rank sum test will be used to compare the differences between the two groups. Multiple comparison correction might be used for p-values to address the multiple testing issues due to measurements at multiple time points.
Time Frame: changes in platelets from pre-op to post-op level, 6 months
Measure: Mean (Standard Deviation); unit: 10e3 platelets/mm^3
Arm/Group | Arm A-Tranexamic Acid | Arm B-Placebo | TXAKIDS
Number analyzed (Participants) | 6 | 6 | 12
10e3 platelets/mm^3
  Platelets (intra-op) | 227.00 (98.04) | 239.84 (75.99) | 233.42 (83.90)
  Platelets (post-op) | 162.33 (25.74) | 168.83 (73.20) | 165.58 (52.42)
Statistical Analysis 1: Comparison: Arm A-Tranexamic Acid vs Arm B-Placebo; Test type: Equivalence — Two-sided test at 0.05 level; p = 0.4286, Wilcoxon rank sum test

3. Secondary Outcome: To Evaluate Changes in Hemoglobin From Pre-op to Post-op Level for Patients Randomized to Receive Perioperative TXA Versus Placebo.
Description: Summary statistics will be provided for the decline in hemoglobin from pre-op to post-op level, for both the TXA and placebo group. Two sample t-test or Wilcoxon rank sum test will be used to compare the differences between the two groups. Multiple comparison correction might be used for p-values to address the multiple testing issues due to measurements at multiple time points.
Time Frame: changes in hemoglobin from pre-op to post-op level, 6 months
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Arm A-Tranexamic Acid | Arm B-Placebo | TXAKIDS
Number analyzed (Participants) | 6 | 6 | 12
g/dL
  Hemoglobin (intra-op) | 11.70 (2.13) | 11.00 (1.64) | 11.35 (1.85)
  Hemoglobin (post-op) | 8.23 (1.30) | 7.77 (0.70) | 8.00 (1.02)
Statistical Analysis 1: Comparison: Arm A-Tranexamic Acid vs Arm B-Placebo; Test type: Equivalence — Two-sided test at 0.05 level; p = 0.9307, Wilcoxon rank sum test

4. Secondary Outcome: To Evaluate Differences in Post-operative Daily Surgical Drain Output for Patients Randomized to Receive Perioperative TXA Versus Placebo.
Description: Summary statistics will be provided for postoperative daily surgical drain output (in milliliters per 24 hour period for the duration of the drain) for each group. The group difference will be compared using two-sample t-test or Wilcoxon rank sum test depending on the distribution of the observed data. Multiple comparison correction might be used for p-values to address the multiple testing issues due to measurements at multiple time points.
Time Frame: Conclusion of surgery to time of drain removal (prior to discharge from inpatient)
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | Arm A-Tranexamic Acid | Arm B-Placebo | TXAKIDS
Number analyzed (Participants) | 6 | 6 | 12
ml | 246.00 (146.81) | 83.20 (79.43) | 144.25 (129.86)
Statistical Analysis 1: Comparison: Arm A-Tranexamic Acid vs Arm B-Placebo; Test type: Equivalence — Two-sided test at 0.05 level; p = 0.0714, Wilcoxon rank sum test

5. Secondary Outcome: To Evaluate Changes in Estimated Blood Loss (EBL) for Patients Randomized to Receive Perioperative TXA Versus Placebo.
Description: The EBL for pre-op to post-op level, for both the TXA treated group and placebo group will be estimated with a two-sided 95% confidence interval. The EBL of the two groups (TXA vs. Placebo) will be evaluated using a two-sample t-test or Wilcoxon rank sum test depending on the distribution of the observed data.
Time Frame: At conclusion of surgery
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | Arm A-Tranexamic Acid | Arm B-Placebo | TXAKIDS
Number analyzed (Participants) | 6 | 6 | 12
ml | 669.67 (551.15) | 808.67 (607.53) | 739.17 (557.78)
Statistical Analysis 1: Comparison: Arm A-Tranexamic Acid vs Arm B-Placebo; Test type: Equivalence — Two-sided test at 0.05 level; p = 0.9004, Wilcoxon rank sum test

6. Secondary Outcome: To Evaluate Log Transfused Blood Volume Between the intra-or Post-operatively for Patients Randomized to Receive Perioperative TXA and Placebo, Respectively.
Description: Mean and Standard Deviation of log Transfused Blood Volume for both the TXA treated group and placebo group will be estimated.
Time Frame: At conclusion of surgery
Measure: Mean (Standard Deviation); unit: log(mL/kg)
Arm/Group | Arm A-Tranexamic Acid | Arm B-Placebo | TXAKIDS
Number analyzed (Participants) | 6 | 6 | 12
log(mL/kg) | 1.68 (0.32) | 1.67 (0.38) | 1.68 (0.34)

7. Secondary Outcome: To Evaluate Log Estimated Blood Loss (EBL) Between the intra-or Post-operatively for Patients Randomized to Receive Perioperative TXA and Placebo, Respectively.
Description: Mean and Standard Deviation of log Estimated Blood Loss for both the TXA treated group and placebo group will be estimated.
Time Frame: At conclusion of surgery
Measure: Mean (Standard Deviation); unit: log(mL)
Arm/Group | Arm A-Tranexamic Acid | Arm B-Placebo | TXAKIDS
Number analyzed (Participants) | 6 | 6 | 12
log(mL) | 6.11 (0.67) | 6.77 (0.56) | 6.38 (0.70)

8. Secondary Outcome: To Evaluate the Association Between the intra-or Post-operatively Transfused Blood Volume and Estimated Blood Loss (EBL) for Patients Randomized to Receive Perioperative TXA and Placebo, Respectively.
Description: Regression model will be used to access the correlation between the log transformed intra-or post-operatively transfused blood volume and EBL.
Time Frame: At conclusion of surgery
Measure: Number; unit: correlation coefficient
Arm/Group | Arm A-Tranexamic Acid | Arm B-Placebo | TXAKIDS
Number analyzed (Participants) | 6 | 6 | 12
correlation coefficient | 0.36 | -0.42 | 0.03

ADVERSE EVENTS:
Time Frame: Adverse events were collected from Post-Anesthesia Care Unit (PACU) to 6 months.
Arm/Group | Arm A-Tranexamic Acid | Arm B-Placebo
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 1/6 | 1/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A-Tranexamic Acid (N=6) | Arm B-Placebo (N=6)
Injury, poisoning and procedural complications - Other (Injury, poisoning and procedural complications) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-06-30): https://cdn.clinicaltrials.gov/large-docs/42/NCT04410042/Prot_SAP_001.pdf
  • Informed Consent Form (2023-06-30): https://cdn.clinicaltrials.gov/large-docs/42/NCT04410042/ICF_000.pdf